CLINICAL TRIAL: NCT06995807
Title: Enhancing the Efficacy of Depression and Low Mood Treatment: A Novel Adjunctive Approach
Brief Title: EL-SHIN Therapy for Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MonashUMalaysia
Record Dates: First submitted 2025-05-07; First posted 2025-05-30 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either continue standard treatment with a control activity (Group A) or receive EL-SHIN® Therapy alongside their usual care (Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EL-SHIN THERAPY (CONTROL GROUP A) (No Intervention): Control Group
- EL-SHIN THERAPY (GROUP B) (Experimental): Group receiving intervention
  Interventions: Other: EL-SHIN THERAPY

INTERVENTIONS:
Other: EL-SHIN THERAPY — Participants will be randomly assigned to Group A and Group B. Group A : Attend a talk on Malaysia Tourism + current coping strategies.
  Group B : EL-SHIN® Therapy + current coping strategies. Duration of therapies: 2 weeks Assessments using (i) DASS-21 (ii) MHQoL (iii) SLEEP QUALITY SCALE (SQS) at baseline, after 1st week & 2nd weeks for both groups. Assessment will be done on end of 3rd week to see effect when EL-SHIN Therapy Stopped.
  Group B participants: Attend a workshop on administration of EL-SHIN® Therapy. Will reinitiate EL-SHIN Therapy on the 4th week and assess on the 8th day to see the effect.
  Arms: EL-SHIN THERAPY (GROUP B)

SUMMARY:
This is a research aiming to find the effectiveness of an innovative therapy, EL-SHIN THERAPY, in ameliorating depressive symptoms.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of EL-SHIN® Therapy, a novel adjunctive intervention in alleviating depressive symptoms.

There are three components in this therapy:

1. Lavender Therapy
2. GRATEFULNESS® Therapy
3. Fasting with exercise and light therapy

The study includes two phases: a quantitative clinical trial and a qualitative focus group.

Assessments will use DASS-21, MHQoL, and SQS scales with the intervention delivered in English over 3-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: Above 18 yrs old
* DASS-21 scores:

"Moderately Depressed (Score: 14-20)", "Moderately Anxious (Score: 10-14)" & "Moderately Stressed (Score: 19-25)"

* Non-Muslim (Due to legal restriction in Malaysia for this religion)
* English literate
* Believers in Creationism

Exclusion Criteria:

* Muslim (legal restrictions in Malaysia for this religion).
* Non-English literate (research will be conducted in English only).
* Individuals with any other medical conditions or on current medication To reduce potential complications or confounding factors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, Female, Non-Binary, Others (to be specified)
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
DASS-21 Scale | 3 to 4 weeks
  Measuring severity of Depression, Anxiety and Stress Level. Higher score indicating more severity in experiencing these symptoms
Mental Health Quality of Life (MHQoL) | 3 to 4 weeks
  Measuring quality of life of individuals. Higher score indicating better quality of life.
Sleep Quality Scale (SQS) | 3 to 4 weeks
  Measuring Sleep Quality of Individuals with higher score denoting more acute sleep problem

CONTACTS AND LOCATIONS:
Overall Officials: AI SHIN LIM, PHD, Principal Investigator — Monash University Malaysia
Locations (1):
- Monash University Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No